CLINICAL TRIAL: NCT01062737
Title: Evaluation of the Structure-modifying Effect and Safety of Avocado-Soybean Unsaponifiable (Piascledine 300) in Hip Osteoarthritis (OA) a 3 Years Multicenter Randomized, Double Blind, Placebo Controlled Trial
Brief Title: Evaluation of the Structure Modifying Effect of Avocado-Soybean Unsaponifiables in Hip Osteoarthritis
Acronym: ERADIAS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Laboratoires Expanscience S.A. (Industry)
Responsible Party: Pr Michel Lequesne, Principal investigator
Other Study IDs: PR 2898
Record Dates: First submitted 2010-02-03; First posted 2010-02-04 (Estimated); Last update posted 2010-02-04 (Estimated); Status verified 2010-02

CONDITIONS: Hip Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Hip

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ASU (Avocado Soybean Unsaponifiable) (Experimental)
  Interventions: Drug: ASU

INTERVENTIONS:
Drug: ASU

SUMMARY:
This study aims to assess the long term (three years) ability of ASU (Avocado Soya unsaponifiable) to slow the decrease of radiographic JSW (Joint Space Width) in hip osteoarthritis (OA). This is a randomized, double blind, comparative, parallel group study versus placebo.

DETAILED DESCRIPTION:
Inclusion criteria:

Primary hip OA, fulfilling ACR criteria, patient over 45 y, painful > 1 year, Lequesne's index > or equal to 3, with minimum JSW at the target hip > 1 mm and < 4 mm on pelvic radiograph.

Primary criterion of efficacy:

The main criterion of efficacy is the change of JSW between baseline and end point. JSW is measured on the narrowest joint on pelvic or target hip X ray by blinded reader.

Randomisation is stratified according JSW at baseline (< 2,5 mm or > or equal to 2,5 mm).

Statistical analysis:

The Full Analysis Set (FAS) is defined by patients with at least one baseline value and one post baseline value.

The main analysis is scheduled on FAS using a Missing At Random (MAR)with a multiple model repeated measure (MMRM)to take in account missing value.

SAP (Statistical Analysis Plan) schedule to analyse JSW change as quantitative variable using an ANCOVA and as qualitative variable (progressors defined as JSW loss upper than 0,5 mm) using Mantel Haentzel test.

ELIGIBILITY:
Inclusion Criteria:

* primary OA of hip,
* ACR criteria,
* older than 45 years,
* symptomatic painful > 1 an,
* Lequesne's index > or equal to 3,
* JSW between 1 and 4 mm on pelvic radiograph.

Exclusion Criteria:

* secondary OA.

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1999-12; Primary Completion 2006-09 (Actual); Study Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
The main criterion of efficacy is the change of JSW between baseline and end point. JSW is measured on the narrowest joint on pelvic or target hip X ray by blinded reader.

CONTACTS AND LOCATIONS:
Locations (1):
- Multiple locations, Paris, France

REFERENCES:
- [Derived] Maheu E, Cadet C, Marty M, Moyse D, Kerloch I, Coste P, Dougados M, Mazieres B, Spector TD, Halhol H, Grouin JM, Lequesne M. Randomised, controlled trial of avocado-soybean unsaponifiable (Piascledine) effect on structure modification in hip osteoarthritis: the ERADIAS study. Ann Rheum Dis. 2014 Feb;73(2):376-84. doi: 10.1136/annrheumdis-2012-202485. Epub 2013 Jan 23. PMID 23345601